CLINICAL TRIAL: NCT06312319
Title: Effects of a Home-based Respiratory Muscle Training on Swallowing Function in Patients With Chronic Stroke
Brief Title: Home-based Respiratory Training on Swallowing in Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Irene Cabrera Martos, Profesor titular de Universidad, Universidad de Granada
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DF0001
Record Dates: First submitted 2024-01-31; First posted 2024-03-15 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Respiratory training added to orofacial exercises (Experimental): Home-based respiratory training of the inspiratory and expiratory muscles using a device added to standard treatment including orofacial exercises.
  Interventions: Device: Respiratory training; Other: Orofacial exercises
- Orofacial exercises (Active Comparator): Standard treatment including orofacial exercises.
  Interventions: Other: Orofacial exercises

INTERVENTIONS:
Device: Respiratory training — Respiratory training using the EMST 150 device to increase inspiratory and expiratory muscle strength.
  Arms: Respiratory training added to orofacial exercises
Other: Orofacial exercises — The exercises will include activities to improve orofacial structures such as mobility, strength and coordination.

SUMMARY:
The aim of this study is to evaluate the effects of a home-based respiratory muscle training on swallowing function in patients with chronic stroke. The patients will be included in a experimental or a control group. The patients in the experimental group will receive a home-based respiratory training using respiratory devices added to standard treatment, while the participants in the control group will only receive the standard treatment.

DETAILED DESCRIPTION:
This study aims to evaluate the effects of a home-based respiratory muscle training on swallowing function in patients with chronic stroke. The patients will be included in a experimental or a control group. The patients in the experimental group will receive home-based respiratory training using respiratory devices added to standard treatment, while the participants in the control group will only receive the standard treatment. The swallowing function will be assessed using specific tools and questionnaires. Secondary outcomes will evaluate the respiratory function. The intervention will have a duration of 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of stroke
* 18 years of age or more

Exclusion Criteria:

* Cognitive impairment or aphasia that prevents the understanding of instructions.
* Tracheostomy.
* Presence of cancer.
* Patients who present another disease of the central nervous system
* Absence of neuromotor competence to carry out the respiratory function tests.
* Central apnea.
* Hypoventilation-obesity syndrome.
* Severe cardiorespiratory impairment (hemodynamic instability, pulmonary embolism, recent pneumonothorax, acute hemoptysis, active respiratory infections, recent myocardial infarction, unstable angina, pulmonary hypertension, uncontrolled asthma, or severe chronic obstructive pulmonary disease).
* Patients with recent otorhinolaryngological, abdominal, or thoracic surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-08-20 (Actual); Primary Completion 2024-03-20 (Estimated); Study Completion 2024-06-20 (Estimated)

PRIMARY OUTCOMES:
Gugging Swallowing screen | Baseline, 6 weeks
  Screening test that indicates the need to evaluate the presence of dysphagia. The scores ranges from 0 to 20, with higher scores indicating better performance. Twenty points are the highest score that a patient can attain, and it means normal swallowing ability without aspiration risk.
Swallowing quality of life questionnaire | Baseline, 6 weeks
  Questionnaire evaluating the impact of swallowing deficits on daily living. The scores range from 0 to 100 metric, with a lower score indicating less quality of life.
cough peak flow | Baseline, 6 weeks
  Evaluation of the strength of cough using a peak flow meter

SECONDARY OUTCOMES:
Forced vital capacity | Baseline, 6 weeks
  This is the maximum amount of air you can forcibly exhale from your lungs after fully inhaling
Forced expiratory volumen in the first second | Baseline, 6 weeks
  refers to the volume of air that an individual can exhale during a forced breath in the first second.
FEV1/FVC ratio | Baseline, 6 weeks
  This is the ratio of the forced expiratory volume in the first one second to the forced vital capacity of the lungs
Respiratory Pressure Meter | Baseline, 6 weeks
  This measure will include the maximal inspiratory and maximal expiratory measures evaluated using a device

CONTACTS AND LOCATIONS:
Overall Officials: Irene Cabrera Martos, Principal Investigator — UGR
Locations (1):
- Faculty of Health Sciences, Granada, Spain